CLINICAL TRIAL: NCT04331730
Title: A Double-Masked, Placebo-Controlled, Dose Ranging Study to Evaluate the Efficacy of Oral AKST4290 With Loading Doses of Aflibercept in Patients With Newly Diagnosed Neovascular Age-Related Macular Degeneration
Brief Title: A Study to Assess the Efficacy and Safety of AKST4290 With Aflibercept in Patients With Newly Diagnosed nAMD
Acronym: PHTHALO-205
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AKST4290-205
Record Dates: First submitted 2020-03-16; First posted 2020-04-02 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AKST4290 (800 mg) + Aflibercept (Experimental): Subjects will receive 400 mg AKST4290 twice daily for 36 weeks, in combination with intravitreal aflibercept injection treatment
  Interventions: Drug: AKST4290; Drug: Aflibercept
- AKST4290 (1600 mg) + Aflibercept (Experimental): Subjects will receive 800 mg AKST4290 twice daily for 36 weeks, in combination with intravitreal aflibercept injection treatment
  Interventions: Drug: AKST4290; Drug: Aflibercept
- Placebo + Aflibercept (Placebo Comparator): Subjects will receive placebo for 36 weeks, in combination with intravitreal aflibercept injection treatment
  Interventions: Drug: Placebo; Drug: Aflibercept

INTERVENTIONS:
Drug: AKST4290 — Oral AKST4290
  Arms: AKST4290 (1600 mg) + Aflibercept; AKST4290 (800 mg) + Aflibercept
Drug: Placebo — Oral placebo
  Arms: Placebo + Aflibercept
Drug: Aflibercept — Aflibercept intravitreal injection

SUMMARY:
This study will evaluate the efficacy and safety of AKST4290 in combination with aflibercept injections in subjects with newly diagnosed neovascular age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
This is a randomized, double-masked, placebo-controlled, dose-ranging, multicenter study to assess the efficacy and safety of AKST4290 administered orally at 400 mg b.i.d. or 800 mg b.i.d. in combination with intravitreal aflibercept injections (IAI), in subjects with newly diagnosed neovascular age-related macular degeneration (nAMD) who are naïve to treatment with anti-vascular endothelial growth factor (anti-VEGF) medications in the study eye. Subjects will be treated with AKST4290 800 mg daily, 1600 mg daily, or placebo for a total of 36 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women with newly diagnosed active Choroidal Neovascularization (CNV) secondary to Age-Related Macular Degeneration (AMD), diagnosed by a retinal specialist with all the following characteristics and ophthalmic inclusion criteria applied to the study eye, as assessed by a central reader:

  * Has been examined by a retinal specialist and found to be eligible to receive Intravitreal Aflibercept Injection (IAI) in the study eye.
  * No prior treatment for Neovascular Age-Related Macular Degeneration (nAMD) in the study eye.
  * Study eye has not undergone pars plana vitrectomy or glaucoma filtering surgery.
  * Participation in studies of investigational drugs must have been discontinued within 30 days or 5 half-lives of the drug (whichever was longer) prior to screening.
  * Central subfield thickness (CST) thickness ≥ 250 microns on SD-OCT (spectral domain OCT) (exclusive of subretinal pigment epithelial fluid, inclusive of SRF).
  * Presence of SRF (subretinal fluid) and/or IRF (intraretinal fluid) on SD-OCT.
  * Total lesion size not greater than 12 disc areas (30.48 mm2) (1 disc area = 2.54 mm2) on FA (fluorescein angiography).
  * If present, subretinal hemorrhage must comprise < 50% of the total lesion area on FA, SD-OCT, or FP/FAF (fundus photography/fundus autofluorescence).
  * No subfoveal fibrosis or atrophy on FA, SD-OCT, or FP/FAF.
  * Active CNV (choroidal neovascularization) membranes with subfoveal leakage or juxtafoveal leakage too close for laser photocoagulation.
* BCVA (Best Corrected Visual Acuity) in the study eye between 70 and 24 letters inclusive.
* Body mass index (BMI) between (and inclusive of) 18 and 40 at screening.

Key Exclusion Criteria:

* Participation in studies of investigational drugs within 30 days or 5 half-lives of the drug (whichever was longer) prior to screening.
* Known hypersensitivity to the active substance or any of the excipients of AKST4290 or aflibercept.
* Active or suspected ocular or periocular infection and/or active, severe intraocular inflammation.
* Any form of macular degeneration that is not age-related (e.g., Best's disease, Stargardt's disease, Sorsby's disease).
* Additional disease in the study eye that could compromise BCVA (i.e., uncontrolled glaucoma (IOP >24) with visual field loss, clinically significant diabetic macular edema, history of ischemic optic neuropathy or retinal vascular occlusion, vitreomacular traction, high myopia > 6 diopters, or genetic disorders such as retinitis pigmentosa).
* Presence of RPE (Retinal Pigment Epithelium) tears or rips in the study eye.
* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate visualization with FP/FAF, FA, or SD-OCT.
* Intraocular surgery in the study eye within 3 months prior to screening.
* Aphakia or total absence of the posterior capsule (yttrium aluminum garnet [YAG] laser capsulotomy permitted in an eye with a posterior chamber intraocular lens if performed a minimum of 1 month prior to enrollment) in the study eye.
* Known allergy to fluorescein sodium.
* Significant alcohol or drug abuse within past 2 years.
* Based on ECG (electrocardiogram) reading, subjects with a risk of QT prolongation.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (21):
- United States (3):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Vitreous Associates of FL, St. Petersburg, Florida
  - Sierra Eye Associates, Reno, Nevada
- Germany (3):
  - Internationale Innovative Ophthalmochirurgie GbR, Düsseldorf
  - nordBLICK Augenklinik Bellevue, Kiel
  - Augentagesklinik Rheine, Rheine
- Hungary (5):
  - Jahn Ferenc Dél-pesti Kórház (Jahn Ferenc South-Pest Hospital), Budapest
  - Magyar Honvédség Egészségügyi Központ, Szemészeti Osztály (Medical Centre, Hungarian Defence Forces, Ophthalmology Department), Budapest
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház (Borsod-Abaúj-Zemplén County Hospital and University Teaching Hospital), Miskolc
  - GANGLION Orvosi Központ, Pécs
  - Szegedi Tudományegyetem Általános Orvostudományi Kar, Szent-Györgyi Albert Klinikai Központ, Szemészeti Klinika, (University of Szeged Faculty of Medicine, Albert-Szent Gyorgyi Health Care, Department of Ophthalmology), Szekszárd
- Poland (10):
  - Tęczówka (IRIS), Bialystok
  - Specjalistyczny Ośrodek Okulistyczny Oculomedica (Specialized Eye Center Oculomedica), Bydgoszcz
  - PROVISUS Sp. z o.o., Częstochowa
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Centrum Medyczne Dietla 19 Sp zoo, Krakow
  - Klinika Chirurgii Siatkówki i Ciała Szklistego Medical University in Lublin, Lublin
  - Szpital św. Wojciecha, Poznan
  - ArtOptica Salon Okulistyczno, Suwałki
  - Centrum Medyczne UNO-MED, Tarnów
  - Central Clinical Hospital of the MSWiA, Warsaw

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Started | 36 | 35 | 36
Completed | 36 | 29 | 34
Not Completed | 0 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept | Total
Number analyzed (Participants) | 36 | 35 | 36 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.4 (8.84) | 74.7 (7.42) | 73.8 (9.34) | 75.0 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 21 | 68
  Male | 14 | 10 | 15 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 35 | 35 | 35 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 36 | 35 | 35 | 106
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 5 | 4 | 4 | 13
  United States | 2 | 3 | 2 | 7
  Poland | 29 | 28 | 30 | 87

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) Per the Early Treatment Diabetic Retinopathy Study (ETDRS) Testing Method
Description: Mean change from baseline in Best Corrected Visual Acuity (BCVA) per the Early Treatment Diabetic Retinopathy Study (ETDRS) testing method. BCVA will be assessed using ETDRS charts at 4 meters initial testing distance and assessed in both eyes. Score range is 0 to 93. A higher score indicates better vision.
Time Frame: Baseline to Week 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Number analyzed (Participants) | 36 | 35 | 36
score on a scale | 10.4 (10.26) | 6.7 (7.89) | 13.7 (7.60)

2. Secondary Outcome: Time to PRN Injection (Arms 1 and 2 Only)
Description: Time to first use of intravitreal aflibercept injection, as needed (AKST4290 Arms only). UNITS: weeks.
Time Frame: Baseline to Week 36
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept
Number analyzed (Participants) | 36 | 35
weeks | 20.6 [19.0 to 24.4] | 20.1 [17.0 to 21.7]

3. Secondary Outcome: Median Number of Aflibercept Injections Received Beginning at Week 12
Description: Median number of injections received beginning at Week 12 as a rate. UNITS: number of injections per week from Week 12
Time Frame: Week 12 to Week 36
Population: The number of injections received per week is defined as the number of IAIs received on or after Week 12 (PRN or scheduled injections) divided by (the analysis Week visit date [or EOS date if subject terminates study early] minus date of Week 12 visit plus one, divided by seven). Data reported reflects subjects with available data for those having received injections from week 12.
Measure: Median (Inter-Quartile Range); unit: number of injections per week
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Number analyzed (Participants) | 36 | 34 | 35
number of injections per week | 0.082 [0.041 to 0.124] | 0.083 [0.042 to 0.124] | 0.125 [0.123 to 0.159]

4. Secondary Outcome: Percentage of Subjects With Best Corrected Visual Acuity (BCVA) Change of ≥ 15 Letters
Description: Percentage of subjects with Best Corrected Visual Acuity (BCVA) change of ≥ 15 letters at Week 36.
Time Frame: Baseline to Week 36
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Number analyzed (Participants) | 36 | 35 | 36
percentage of participants | 30.6 [16.3 to 48.1] | 14.3 [4.8 to 30.3] | 41.7 [25.5 to 59.2]

5. Secondary Outcome: Mean Change in Central Subfield Thickness (CST) Compared With Control Through Week 12
Description: Mean change in Central Subfield Thickness (CST) compared with control through Week 12. UNITS: micrometre
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: micrometre
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Number analyzed (Participants) | 36 | 35 | 36
micrometre | -135.3 (122.66) | -162.7 (118.91) | -159.5 (128.00)

6. Secondary Outcome: Number of Participants With Adverse Events Assessed by Intensity
Description: Number of Participants with Adverse Events categorized by intensity
Time Frame: Screening to Week 40
Measure: Count of Participants; unit: Participants
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Number analyzed (Participants) | 36 | 35 | 36
Participants
  Mild TEAE | 15 | 10 | 11
  Moderate TEAE | 8 | 7 | 8
  Severe TEAE | 3 | 9 | 1
  No TEAE | 10 | 9 | 16

7. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) Per the Early Treatment Diabetic Retinopathy Study (ETDRS) Testing Method as Compared With Control
Description: Mean change in Best Corrected Visual Acuity (BCVA) letter score per the Early Treatment Diabetic Retinopathy Study (ETDRS) testing method from Week 12 as compared to control at Week 36. BCVA will be assessed using ETDRS charts at 4 meters initial testing distance and assessed in both eyes. Score range is 0 to 93. A higher score indicates better vision.
Time Frame: Week 12 to Week 36
Population: Reported data follows the pre-specified analyses and tables generated per the Statistical Analysis Plan for additional analyses of the primary endpoint. Change from Week 12 in BCVA ETDRS letters read is reported for the AKST4290 combined group and Placebo and will include a similar REML-based MMRM analysis as described for the primary endpoint; a covariate of letters read at Week 12 will be included in lieu of baseline letters read.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AKST4290 + Aflibercept Pooled (800 mg or 1600 mg): Subjects will receive 400 mg or 800 mg AKST4290 twice daily for 36 weeks, in combination with intravitreal aflibercept injection treatment
  AKST4290: Oral AKST4290
  Aflibercept: Aflibercept intravitreal injection
Arm/Group | AKST4290 + Aflibercept Pooled (800 mg or 1600 mg) | Placebo + Aflibercept
Number analyzed (Participants) | 71 | 36
score on a scale | 1.1 (5.98) | 2.3 (5.35)

8. Secondary Outcome: Time to the First Visit Where PRN Injection Criteria Are Met
Description: Time to the first visit where PRN injection criteria are met starting at Week 12 will be calculated in weeks as the first date where PRN injection criteria are first met minus the date of first dose of study drug plus one, divided by seven. Subjects who do not experience the event of interest (meet the criteria for PRN IAI) while on the study will be censored at their last visit completed through Week 36. Units: weeks
Time Frame: Week 12 to the first visit meeting PRN injection criteria through week 36
Population: Data reflects subjects having received injections from week 12. Subjects who do not experience the event of interest (i.e., receive a PRN injection, meet the criteria for PRN IAI) while on the study were censored at their last visit completed through Week 36, as applicable.
Measure: Median (Full Range); unit: weeks
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
Number analyzed (Participants) | 29 | 31 | 24
weeks | 20.6 [12.9 to 39.0] | 20.1 [12.1 to 37.1] | 20.4 [11.7 to 37.4]

ADVERSE EVENTS:
Time Frame: From Screening through End of Study, approximately 42 weeks
Description: AEs were captured beginning at time of informed consent through EOS. AE status was followed by the investigator until resolved or considered stable, unless the subject was lost to follow up
Arm/Group | AKST4290 (800 mg) + Aflibercept | AKST4290 (1600 mg) + Aflibercept | Placebo + Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 3/36 | 3/35 | 0/36
Other Adverse Events (participants affected / at risk) | 26/36 | 26/35 | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKST4290 (800 mg) + Aflibercept (N=36) | AKST4290 (1600 mg) + Aflibercept (N=35) | Placebo + Aflibercept (N=36)
COVID-19 (Infections and infestations) | 0 | 2 | 0
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AKST4290 (800 mg) + Aflibercept (N=36) | AKST4290 (1600 mg) + Aflibercept (N=35) | Placebo + Aflibercept (N=36)
Electrocardiogram QT prolonged (Investigations) | 5 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Eye pain (Eye disorders) | 3 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
COVID-19 (Infections and infestations) | 0 | 4 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 2
Hepatic enzyme increased (Investigations) | 0 | 3 | 0
Liver function test abnormal (Investigations) | 1 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Product residue present (Investigations) | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Blood pressure increased (Investigations) | 0 | 2 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT04331730/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT04331730/SAP_001.pdf